CLINICAL TRIAL: NCT02626975
Title: MRI Study of Ballooning and Ligamentisation Short Transplants ACL Hamstring According to Technical DT4
Acronym: MRI-DT4
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_50; 2014-A01413-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Deficiency of Anterior Cruciate Ligament; Displacement of Bone Allograft
Keywords: knee; short hamstring autograft; ligament; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACL reconstruction ballooning: ACL reconstruction with short hamstring tendon autograft
  * arm ballooning
  * arm no ballooning

SUMMARY:
MRI study of ballooning and ligamentisation short transplants of anterior cruciate ligament (ACL) according to DT4 technique in 60 patients with more than one year of follow up.

DETAILED DESCRIPTION:
Monocentric study in the CHRU Lille in which the first goal is to estimate the frequency of tunnel's ballooning in a surgical anterior cruciate ligament reconstruction using short transplants of hamstrings.

the secondary goals Secondary goals of this study are the estimation of ligamentisation if ballooning or not, the comparison of sagittal laximetry between "ballooned" group and "not ballooned"one, the clinical results in IKDC score (International Knee Documentation Committee subjective fee form) and KOOS (Knee injury Osteoarthritis Outcome Score) between the "ballooned" group and the "not ballooned"one.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients of both sexes with an hamstring ACL ligamentoplasty done in our institution with a follow up of 1 year
* isolated ACL ligamentoplasty
* insured patients with a signed informed consent

Exclusion Criteria:

* follow up inferior of 1 year
* absolute contraindication to knee MRI
* gadolinium allergy
* severe renal failure
* non isolated ACL ligamentoplasty
* patient under guardianship, minor
* pregnant woman or nursing mother

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with an hamstring ACL ligamentoplasty with a follow up of at least 1 year
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2016-06-23 (Actual); Study Completion 2016-06-23 (Actual)

PRIMARY OUTCOMES:
frequency of balloonisation | 1 year
  oversize of the diameters of femoral and /or tibial tunnels more than 50% of their surgical diameter

SECONDARY OUTCOMES:
frequency of ligamentisation | 1 year
  fixation on MRI of gadolinium in ligament graft
laximetry done with genurob* | 1 year
  measure of the residual anterior laxity on an electronic device
Knee Injury and Osteoarthritis Outcome Score | 1 year
  clinical measures
International Knee Documentation Commitee (IKDC) Score | 1 year
  clinical measures

CONTACTS AND LOCATIONS:
Overall Officials: Gilles PASQUIER, MD, PhD, Study Chair — University Hospital, Lille
Locations (1):
- University Hospital, Hôpital Salengro, Lille, France

IPD SHARING:
Plan to Share IPD: No